CLINICAL TRIAL: NCT06894745
Title: Positron Emission Tomography (PET) Imaging of the Enhanced Permeability and Retention (EPR) Effect With [89Zr]DFO-starPEG in Patients With Solid Tumors
Brief Title: PET [89Zr]DFO-starPEG in Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Flavell, MD, PhD (Other)
Collaborators: ProLynx LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robert Flavell, MD, PhD, Associate Professor in Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25921; 1R01CA266666-01A1 (NIH); NCI-2025-02151 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor; Solid Carcinoma; Soft Tissue Lesion
Keywords: Dosimetry; Imaging
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A: Multiple Scans (89Zr]DFO-starPEG) (Experimental): Participants will be administered a single, intravenous microdose (1 - 2 millicurie (mCi) of [89Zr]DFO-starPEG, followed by whole-body positron emission tomography (PET) imaging. PET imaging will be conducted at the following times after [89Zr]DFO-starPEG administration:
  2 hours (±30 min), 24 (±4) hours (1 day), 48-72 hours (2-3 days), and 120-216 hours (5-9 days).
  Interventions: Drug: 89-zr-dfo-star polyethylene glycol (StarPEG); Procedure: Whole Body Positron Emission Tomography (PET); Procedure: Specimen Collection
- Cohort B: Single Scan (89Zr]DFO-starPEG) (Experimental): Participants will be administered a single, intravenous microdose (1 - 2 mCi) of [89Zr]DFO-starPEG, followed by whole-body PET imaging will be conducted 120-216 hours (5-9 days) after [89Zr]DFO-starPEG administration.
  Interventions: Drug: 89-zr-dfo-star polyethylene glycol (StarPEG); Procedure: Whole Body Positron Emission Tomography (PET); Procedure: Specimen Collection

INTERVENTIONS:
Drug: 89-zr-dfo-star polyethylene glycol (StarPEG) — Given intravenously (IV)
  Other Names: [89Zr]DFO-starPEG
Procedure: Whole Body Positron Emission Tomography (PET) — Imaging procedure
  Other Names: Whole Body PET Scan; Whole Body PET
Procedure: Specimen Collection — Urine and blood specimens will be collected for correlative studies
  Other Names: Biospecimen Collection

SUMMARY:
This is a first-in-human, pilot study of the novel PET-imaging radiotracer [89Zr]DFO-starPEG. The study is designed to obtain preliminary data to support future development of this agent as an imaging surrogate to visualize enhanced permeability and retention (EPR)-mediated tracer uptake before administration of EPR-based nanomedicines.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To descriptively report patterns of [89Zr]DFO-starPEG uptake on whole-body PET (Cohorts A & B).

II. To determine the radiation dosimetry following [89Zr]DFO-starPEG administration (Cohort A).

SECONDARY OBJECTIVES:

I. To determine the safety of [89Zr]DFO-starPEG (Cohorts A & B).

EXPLORATORY OBJECTIVES:

I. To study the pharmacokinetics of [89Zr]DFO-starPEG and estimate its half-life (Cohort A).

OUTLINE:

Participants will be assigned to one of 2 cohorts:

* COHORT A: Participants will receive multiple scans over time
* COHORT B: Participants will receive a scan at a single time point

Participants will be followed for adverse events for approximately 1 week after radiotracer administration until the Day 5-9 visit.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmation of solid tumor malignancy.
2. Any solid tumor malignancy, with at least one soft tissue lesion measurable at 1 centimeter (cm) or greater in short axis measurement on cross sectional imaging such as Computerized tomography (CT), Magnetic resonance imaging (MRI), or Positron Emission Tomography (PET)/CT.
3. Clinically able to undergo PET/CT imaging.
4. Age >= 18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 or Karnofsky ≥ 50%.
6. Adequate organ function as defined below within 0-28 days before [89Zr]DFO-starPEG administration:

   * Total bilirubin: ≤ 1.5 x institutional upper limit of normal (ULN) (unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits) .
   * Aspartate aminotransferase (AST)/ serum glutamic-oxaloacetic transaminase (SGOT) ≤ 3 x ULN.
   * Alanine aminotransferase (ALT)/ serum glutamic-pyruvic transaminase (SGPT) ≤ 3 x ULN.
   * Estimated creatinine clearance: ≥ 60 mL/min, calculated using the Cockcroft-Gault equation or 24 hour urine collection.
7. Females of reproductive potential (defined below) must be willing to undergo a urine or serum pregnancy test (i.e., human chorionic gonadotropin test) within 72 hours before administration of [89Zr]DFO-starPEG. A female is considered to NOT be of reproductive potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice), if they meet either of the following two criteria: (1) has reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause); or (2) has undergone surgical sterilization (i.e., hysterectomy and/or bilateral oophorectomy for removal of uterus and/or ovaries). The result of the urine or serum pregnancy test must be negative in order to initiate the [89Zr]DFO-starPEG administration. If a urine pregnancy test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the individual must be excluded from participation if the serum pregnancy result is positive. Pregnant individuals are excluded from this study because there is an unknown but potential risk for adverse effects in the unborn child secondary to treatment of the study participant with [89Zr]DFO-starPEG.
8. Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or endpoints of this study are eligible.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Individuals with a contraindication to PET-CT imaging (e.g., severe claustrophobia).
2. Individuals who are pregnant or breastfeeding/chestfeeding. Pregnant and breastfeeding/chestfeeding individuals are excluded because there is an unknown but potential risk for adverse effects in the unborn/nursing child secondary to treatment of the study participant with [89Zr]DFO-starPEG. Females of childbearing potential must have a negative pregnancy test before administration of [89Zr]DFO-starPEG, as outlined in inclusion criterion #7. Breastfeeding/chestfeeding should be discontinued before administration of [89Zr]DFO-starPEG.
3. Individuals who do not agree to follow the below contraception requirements:

   * Females of reproductive potential (defined below) must agree to use two forms of contraception, consisting of a barrier method (such as condoms) in combination with a secondary complementary method (such as hormonal, intrauterine device (IUD), etc.), or strict abstinence, for the duration of study participation and for 1 month after administration of [89Zr]DFO-starPEG.
   * A female is considered to NOT be of reproductive potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice), if they meet either of the following two criteria: (1) has reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause); or (2) has undergone surgical sterilization (i.e., hysterectomy and/or bilateral oophorectomy for removal of uterus and/or ovaries).
4. Hypersensitivity to [89Zr]DFO-starPEG or any of its excipients.
5. Individuals with any condition or social circumstance that, in the opinion of the investigator, would impair the participant's ability to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Median Maximum Standardized Uptake Value (SUVmax) by cohort | Up to 9 days
  The median and range for intra-tumoral SUVmax within metastatic lesions will be descriptively reported, to assess for intra-tumoral heterogeneity and differences in uptake by site of disease.
Tumor-to-background signal ratio (muscle) | Up to 9 days
  Adjusted SUVmax data will be averaged across up to 15 lesions within a given patient (SUVmax-avg). VOI will also be placed around the aortic blood pool and paraspinal musculature. Tumor to muscle SUV ratios will be calculated by dividing tumoral SUV by muscle SUV, respectively
Tumor-to-background signal ratio (blood) | Up to 9 days
  Adjusted SUVmax data will be averaged across up to 15 lesions within a given patient (SUVmax-avg). VOI will also be placed around the aortic blood pool and paraspinal musculature. Tumor to blood SUV ratios will be calculated by dividing tumoral SUV by blood SUV.
Mean absorbed dose of PET [89Zr]DFO-starPEG (Cohort A) | Up to 9 days
  Volumes of interest (VOIs) will be drawn around regions identified on the scans that exhibits clearly elevated uptake over the background. Time-activity curves will be generated for each organ, and curve-fitting will be performed to derive the time-integrated activity coefficients (TIACs, also known as residence times). TIACs will be entered into the OLINDA software. The results from all participants in the dosimetry cohort will be combined to allow the calculation of mean, standard deviation (SD), and range of radiation-absorbed doses to individual organs as well as effective dose.

SECONDARY OUTCOMES:
Proportion of participants with treatment-emergent adverse events | Up to 9 days
  Adverse events reported after infusion will be graded according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 by cohort will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Flavell, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No